CLINICAL TRIAL: NCT01058070
Title: An Observational Clinical Feasibility Study of the Magnetic Esophageal Sphincter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1306-US, 1030-IT, 1709-NL; NCT01057992 (obsolete NCT alias); NCT01058564 (obsolete NCT alias)
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Implantable Device (Experimental): Subjects who meet eligibility criteria are implanted with the Magnetic Esophageal Sphincter device (MES)
  Interventions: Device: Torax Medical, Inc. LINX Reflux Management System

INTERVENTIONS:
Device: Torax Medical, Inc. LINX Reflux Management System — Implantable device, Magnetic Esophageal Sphincter

SUMMARY:
Magnetic Esophageal Sphincter implant is intended to reinforce Esophageal Sphincter function in the treatment of Gastroesophageal Reflux Disease (GERD)

DETAILED DESCRIPTION:
The purpose of this feasibility study is to collect preliminary performance and safety information and develop procedural optimization for the Torax Medical Inc. Magnetic Esophageal Sphincter device (MES) in reinforcement of Esophageal Sphincter function to treat Gastroesophageal Reflux Disease (GERD). The information from this study will be used to support the design and conduct of an expanded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, < 85 years, life expectancy > 3yrs.
* Documented history of GERD symptoms such as heartburn and/or regurgitation.
* On daily PPI treatment for at least 3-months.
* Responsive to PPI treatment.
* GERD symptoms, in absence of PPI therapy (minimum 10 days).
* Ambulatory Esophageal pH < 4 for ≥ 5% time or pH < 4 for ≥ 3% time in supine position.
* Patient is a surgical candidate.
* Patient is willing and able to cooperate with follow-up examinations.
* Patient has been informed of the study procedures and the treatment and has signed an informed consent form and provided authorization to use and disclose information for research purposes (HIPAA).

Exclusion Criteria:

* The procedure is an emergency procedure.
* Patient is currently being treated with another investigational drug or investigational device.
* Patient has had prior gastric or esophageal surgery.
* Patient has had any previous endoscopic intervention for GERD
* Patient has suspected or confirmed esophageal or gastric cancer.
* Patient has any size paraesophageal hiatal hernia or sliding hiatal hernia ≥3cm. (Investigator to identify and record type of hiatal hernia at the time of assessment (i.e. para-esophageal, sliding)).
* Patient's esophageal motility is less than 35 mmHg peristaltic amplitude on wet swallows or > 30% failed (non-propulsive) peristaltic sequences.
* Patient has esophagitis - Grade B, C, D (LA Classification).
* Patient has Barretts Esophagus.
* Patient has BMI > 35.
* Patient has symptoms of dysphagia or indications of dysphagia from barium esophagram.
* Patient has Scleroderma and/or Achalasia.
* Patient has an esophageal stricture or gross esophageal anatomic abnormalities (obstructive lesions, etc.).
* Patient has an electrical implant or metallic, abdominal implant(s).
* Patient cannot understand trial requirements or is unable to comply with follow-up schedule.
* Patient is pregnant or nursing, or plans to become pregnant.
* Patient has a psychiatric disorder.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2007-02; Primary Completion 2009-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ganz, MD, Principal Investigator — Minnesota Gastroenterolgy, PA
Locations (5):
- United States (3):
  - University of Southern California, Keck School of Medicine, Los Angeles, California
  - Chapman Medical Center, Orange, California
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
- Policlinico San Donato, Milan, Italy
- Academisch Medisch Centrum (AMC), Amsterdam, Netherlands

REFERENCES:
- [Background] Bonavina L, Saino GI, Bona D, Lipham J, Ganz RA, Dunn D, DeMeester T. Magnetic augmentation of the lower esophageal sphincter: results of a feasibility clinical trial. J Gastrointest Surg. 2008 Dec;12(12):2133-40. doi: 10.1007/s11605-008-0698-1. Epub 2008 Oct 10. PMID 18846406
- [Background] Bonavina L, DeMeester T, Fockens P, Dunn D, Saino G, Bona D, Lipham J, Bemelman W, Ganz RA. Laparoscopic sphincter augmentation device eliminates reflux symptoms and normalizes esophageal acid exposure: one- and 2-year results of a feasibility trial. Ann Surg. 2010 Nov;252(5):857-62. doi: 10.1097/SLA.0b013e3181fd879b. PMID 21037442
- [Background] Lipham JC, DeMeester TR, Ganz RA, Bonavina L, Saino G, Dunn DH, Fockens P, Bemelman W. The LINX(R) reflux management system: confirmed safety and efficacy now at 4 years. Surg Endosc. 2012 Oct;26(10):2944-9. doi: 10.1007/s00464-012-2289-1. Epub 2012 Apr 27. PMID 22538694
- [Background] Saino G, Bonavina L, Lipham JC, Dunn D, Ganz RA. Magnetic Sphincter Augmentation for Gastroesophageal Reflux at 5 Years: Final Results of a Pilot Study Show Long-Term Acid Reduction and Symptom Improvement. J Laparoendosc Adv Surg Tech A. 2015 Oct;25(10):787-92. doi: 10.1089/lap.2015.0394. Epub 2015 Oct 5. PMID 26437027

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Implantable Device
Started | 44
Completed | 33
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Implantable Device
Number analyzed (Participants) | 44
Age, Continuous [Mean (Full Range); unit: years] | 42.8 [19.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 26
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 25.7 [19.0 to 38.0]
% time esophageal pH<4 [Mean (Full Range); unit: percentage] — The time during which esophageal pH is less than 4.0 divided by the total recording time expressed in percentage.
  percentage | 11.9 [2.7 to 38.2]
Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) [Mean (Full Range); unit: scores on a scale] — Scoring scale is from 0 to 5 with 0=no symptoms to 5=symptoms are incapacitating. The maximum value score is 50.
  scores on a scale | 26.5 [10.0 to 39.0]

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Incidence of All Adverse Events at Various Time Points.
Time Frame: 5 years
Measure: Number; unit: participants
Groups:
- LINX Study Subjects: Subjects implanted with LINX device
Arm/Group | LINX Study Subjects
Number analyzed (Participants) | 44
participants | 29

2. Primary Outcome: To Monitor the Improvement of GERD Symptoms.
Description: Percentage of participants with a 50% or more reduction in total GERD-HRQL score is indicative of a substantial improvement in GERD symptoms
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Implantable Device
Number analyzed (Participants) | 33
percentage of participants | 93.9

ADVERSE EVENTS:
Time Frame: Pre-discharge, 2-Weeks, 6-Weeks, 3-Months, 6-Months, 12-Months, 18-Months, 24-Months, 30-Months, 36-Months, 42-Months, 48-Months, 54-Months, and 60-Months Follow-up
Description: An adverse event (AE) is any undesirable/unusual experience that occurs to a subject during the clinical study, whether or not considered device related, including, (but not limited to) those events that result from the use as stipulated in the protocol.
Arm/Group | Implantable Device
Serious Adverse Events (participants affected / at risk) | 3/44
Other Adverse Events (participants affected / at risk) | 25/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implantable Device (N=44)
Vomiting & Nausea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Chest Pain (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Implantable Device (N=44)
Dysphagia (Gastrointestinal disorders) | 20
Vomiting & Nausea (Gastrointestinal disorders) | 1
Pain (General disorders) | 3
Device explant/reoperation (Surgical and medical procedures) | 1
Stomach bloating (Gastrointestinal disorders) | 2
No improvement (General disorders) | 3
Inability to belch or vomit (Gastrointestinal disorders) | 2
Heartburn (Gastrointestinal disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other